CLINICAL TRIAL: NCT02170753
Title: Regional Manual Therapy and Motor Control Exercise for the Management of Chronic Low Back Pain With Hip and Spine Motion Loss: A Randomized Clinical Trial
Brief Title: Regional Manual Therapy and Motor Control Exercise for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Texas Physical Therapy Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 042014-066
Record Dates: First submitted 2014-06-18; First posted 2014-06-23 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Low Back Pain; Musculoskeletal Pain
MeSH Terms: conditions — Low Back Pain; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regional manual therapy (Experimental): The experimental group will receive regional thoracic, pelvic, and hip manual therapy and a standard physical therapy approach including motor control exercise and local lumbar spine manual therapy
  Interventions: Procedure: Regional manual therapy; Procedure: Standard physical therapy
- Standard physical therapy (Active Comparator): The control group will receive standard physical therapy including motor control exercise and local lumbar spine manual therapy.
  Interventions: Procedure: Standard physical therapy

INTERVENTIONS:
Procedure: Regional manual therapy — The experimental group will receive regional thoracic, pelvic, and hip manual therapy and a standard physical therapy approach including motor control exercise and local lumbar spine manual therapy.
  Arms: Regional manual therapy
Procedure: Standard physical therapy — The control group will receive standard physical therapy including motor control exercise and local lumbar spine manual therapy.

SUMMARY:
Purpose: The primary purpose of this study is to determine whether or not the addition of thoracic, pelvic, and hip manual therapy to a standard physical therapy (PT) approach consisting of motor control exercises and lumbar spine manual therapy is better than standard PT alone at improving thoracolumbar spine range of motion (ROM), hip ROM, pain intensity, disability level, and perceived change in patients with chronic low back pain (CLBP) and movement coordination impairments.

Hypothesis: In a CLBP subgroup with movement coordination impairments, participants receiving thoracic, pelvic, and hip manual therapy with standard PT will be superior to participants receiving standard PT alone at improving thoracolumbar spine ROM, hip ROM, pain intensity, physical disability level, and perceived change at two, four, and 12 weeks after initiating treatment.

DETAILED DESCRIPTION:
This study will use a 2x4 factorial mixed design with a between-factor independent variable (IV) of group and a within-factor IV of time. The dependent variables include hip ROM, segmental mobility of the thoracolumbar spine, pain, disability level, and patients' perceived rating of change (GROC). Hip ROM and spinal mobility variables will be measured by the researchers, while pain, disability level, and GROC score will be measured by self-reported questionnaires.

The experimental group will receive a motor control exercise program and manual therapy to the hips and spine corresponding to the individual's unique mobility impairments. The comparison group will receive a motor control exercise program and manual therapy to the lumbar spine only. Both groups will receive treatments at an outpatient clinic 2 times a week for 4 weeks. All outcome measures will be collected at baseline (except the GROC), and then at two weeks, four weeks, and twelve weeks after beginning treatment.

All study participants will receive a motor control exercise program consistent with standard of care. Exercises will be targeted to the abdominals, hip flexors, back extensors, hip extensors, hip flexors, hip abductors, and hip adductors, but will begin with those muscles that test weakest in the clinical exam. Generally, exercises for each subject begin with isolated isometric contractions to ensure adequate motor control, and progress through various degrees of agonist loading with co-contraction of synergists using isotonic open or closed chain movements. Instructions to gradually increase time under tension to a maximum of 30 seconds for four repetitions will be used in order to provide an element of graded-activity exposure and to reflect the tonic nature of stabilizing muscles. Participants unable to complete all exercises by the end of the fourth week will be instructed on how to progress to the final exercises with their independent home exercise program.

In addition to a motor control exercise program, all participants will receive manual therapy to the lumbar spine. Standard PT manual therapy will be limited to non-thrust passive accessory (PA) mobilizations from L1-L5 or soft tissue mobilization to the lumbar paraspinals or quadratus lumborum. Only the participants in the experimental group will receive manual therapy to the hips and thoracic spine according to the mobility impairments identified during the initial testing session. The manual therapy interventions utilized at the hips and thoracic spine are considered standard of care for treatment of those regions, but could be considered experimental for treatment of low back pain. Regional manual therapy will include a variety of thrust and non-thrust techniques targeting the thoracic, lumbopelvic, or hip joints. Hip-based techniques including anterior-posterior hip mobilization, caudal thrust or non-thrust mobilization, and posterior-to-anterior mobilization will be performed. The choice of initiating or suspending a specific manual therapy technique and the grade of treatment will be left to the discretion of the treating therapist (other than the PI). Prior to the commencement of the study, all treating physical therapists will be trained in administration of standard motor control exercises and manual therapy.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 65
* have an active complaint of non-specific low back pain for at least three months
* demonstrate hypomobility of the thoracic or lumbar regions on at least one spinal level
* demonstrate at least two of the following unilateral or bilateral hip ROM deficits: hip flexion < 110°, hip extension loss > 6°, or hip rotation < 30° internally or externally
* demonstrate any one of the following: pain that worsens with sustained end- range movements or positions, lumbar hypermobility, diminished trunk or pelvic muscle strength and endurance, or movement coordination impairments during community/work activities
* Modified Oswestry Score ≥ 30%

Exclusion Criteria:

* evidence of red flags, including fracture, infection, spinal tumor, or cauda equina syndrome
* pain that can be centralized through repeated movements
* signs of hyporeflexia, hypoesthesia, and myotomal weakness indicative of nerve root compression
* pregnancy
* systemic inflammatory conditions such as rheumatoid arthritis or ankylosing spondylitis
* inability to safely tolerate manual therapy to the spine or hips
* injections to the low back within the 2 weeks preceding the initial evaluation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Disability level | Baseline and 2 weeks, 4 weeks, and 12 weeks after beginning treatment
  A subjective report of the participant's average level of perceived disability with functional tasks due to LBP as measured by the Modified Oswestry Low Back Pain Disability Questionnaire (ODQ).

SECONDARY OUTCOMES:
Change in Thoracolumbar spine range of motion | Baseline and 2 weeks, 4 weeks, and 12 weeks after beginning treatment
  Testing for this study will be performed using the Valedo Shape, which is a wheeled skin-surface device containing accelerometers that record inter-segmental distance and change of inclination of spinous processes.
Change in Hip range of motion | Baseline and 2 weeks, 4 weeks, and 12 weeks after beginning treatment
  An inclinometer will be used to measure hip range of motion in the sagittal and transverse planes as measured in degrees.
Change in Pain intensity | Baseline and 2 weeks, 4 weeks, and 12 weeks after beginning treatment
  A subjective report of the participant's average low back pain intensity over the previous 24 hours as measured by the Numeric Pain Rating Scale (NPRS).
Change in Perceived change | 2 weeks, 4 weeks, and 12 weeks after beginning treatment
  A subjective report of the participant's perceived level of improvement from the point that they began treatment as measured by the Global Rating of Change (GROC) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Zafereo, MPT, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Health Professions Physical Therapy Clinic, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No